CLINICAL TRIAL: NCT01513603
Title: Phase II Trial of CLAG-M in Relapsed ALL
Brief Title: Trial of Cladribine, Cytarabine, Mitoxantrone, Filgrastim (CLAG-M) in Relapsed Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Karen Seiter, Professor of Medicine, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-10,442
Record Dates: First submitted 2012-01-11; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Burkitts Leukemia/Lymphoma; Chronic Myelogenous Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cladribine; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLAG-M (Experimental)
  Interventions: Drug: CLAG-M

INTERVENTIONS:
Drug: CLAG-M — IV times 5 days
  Other Names: Leustatin; Ara-C; Novantrone
Drug: CLAG-M — Chemotherapy
  Other Names: Cladribine (Leustatin); Cytarabine (Ara-c); Mitoxantrone (Novantrone)

SUMMARY:
CLAG-M is an active, well tolerated regimen in acute myelogenous leukemia. Each of the agents is active in Acute Lymphoblastic Leukemia (ALL) as well. The current trial will determine the efficacy of the regimen in patients with relapsed ALL.

DETAILED DESCRIPTION:
Patients will receive standard dose CLAG-M (cladribine, cytarabine, mitoxantrone, filgrastim). Standard support care will be given. Efficacy will be assessed through bone marrow examinations and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute lymphoblastic leukemia,
* Burkitts leukemia/lymphoma,
* Lymphoid blastic CML,
* Lymphoblastic lymphoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission percentage | 1 month

SECONDARY OUTCOMES:
Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Seiter, MD, Principal Investigator — New York Medical College
Locations (1):
- Westchester Medical Center/New York Medical College, Valhalla, New York, United States